CLINICAL TRIAL: NCT05103267
Title: Tauropace Reduces Infection After Cardiac Electronic Implantable Device Implantation in Heart Failure Patients
Brief Title: Tauropace to Prevent Cardiac Implantable Device Infections in Heart Failure Patients
Acronym: TRICE-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Rapacciuolo, Principal Investigator, Clinical Professor, Federico II University
Other Study IDs: 01102101
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Infection Cardiac; Heart Failure; Cardiac Implantable Electronic Device Infections; High Risk
Keywords: cardiac implantable electronic device infection
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tauropace in high risk participants: TauroPace™ is a CE marked (certified) medical device defined as a "Disinfecting Solution to Eradicate Airborne Microbial Contamination on the Surface of Cardiac Impiantable Electronic Devices (CIED)".
  TauroPace™ is to eradicate environmental microbial contamination on the surface of any CIED during implantation or revision procedure.
  TauroPace™ is intended to be used during CIED surgery procedure in any adult participant at high risk of CIED infections
  Interventions: Device: Tauropace

INTERVENTIONS:
Device: Tauropace — TauroPace™ contains disinfecting substances to eradicate environmental microbial contamination on the surface of cardiac implantable electronic devices (CIEDs). The surface of the CIED is moistened with TauroPace™ during the implantation procedure to create a hostile environment on the surface of the CIED.

SUMMARY:
The main purpose of the study is to evaluate the ability of the Tauropace to reduce major cardiac implantable electronic device (CIED) infections through 12-months post-procedure following CIED in heart failure participants. The secondary endpoint is to prospectively characterize the performance of Tauropace in participants whose CIED system includes a transvenous RV defibrillation lead.

DETAILED DESCRIPTION:
TRICE-HF is a prospective, multi-center, post-market, interventional clinical study. The main purpose of the study is to evaluate the ability of the Tauropace to reduce major CIED infections through 12-months post-procedure following CIED in heart failure patients. The secondary endpoint is to prospectively characterize the performance of Tauropace in subjects whose CIED system includes a transvenous RV defibrillation lead. These features include the lead integrity alert (LIA), lead noise alert (LNA), RV pacing impedance, and high voltage (HV) pacing impedance to detect events that affect a RV lead's pacing, sensing, or defibrillation circuit lead system events (LSE).

The study will be conducted at up to 10 sites in Italy with up to 500 subjects enrolled.

The enrollment period is expected to start in November 2021 and to take approximately 12 months. Participants will be followed for a minimum of 12 months. Therefore, the anticipated study duration is approximately 24 months and subjects may be followed for up to 24 months depending on when they enroll in the study.

This study is a nonrandomized registry; hence no formal control group will be used. In order to compare our follow-up data, the investigators performed an electronic search of the PubMed and Embase, including all RCTs, retrospective or prospective studied that resulted in CIED infection rates.

The investigators excluded all studies that included patients with abdominal device implants.

No restrictions were imposed on the sample size of the studies. Incidence CIED infections rate or Odds Ratio with 95% confidence intervals were presented as a summary statistic, with the use of the random effects model postulated by DerSimonian and Laird.

Meta-regression was performed to assess the relationship between the magnitude of the treatment effect and different predictors. To estimate the CIED infections incidence in subgroups with certain risk factors, the investigators used the percentage of patients with diabetes, chronic renal failure, undergoing replacement/upgrade/revision procedure, and other CIED infections risk factors, as continuous variables. The investigators predicted a percentage of diabetes and Chronic renal failure patients in our population of 20% and 45 % respectively, but will be able to modify the comparison parameters based on the real percentage of risk factors in the enrolled participants.

Statistical analysis was performed using the "meta" package, with "metagen", "metabin" and "metareg" command, in R programming, R version 4.0.2 (2020-06-22). Results were considered statistically significant if the 2-sided P<0,05.

A 2-sample, 1-sided Fischer Exact test will be used to test the primary efficacy endpoint versus the benchmark rate.

Baseline characteristics will be compared using a Student t test for continuous variables or a Fisher's exact/chi-square test for categorical variables. A Fisher's exact test will be used for sparse data (i.e., np <5 or nq <5). CIED infection and mechanical complication data among ICD and CRT subjects will be compared using the chi-square or Fisher's exact tests. A Fisher's exact test will be used for sparse data.

The study may be considered successful at the first analysis in which the primary objective is met.

ELIGIBILITY:
Inclusion Criteria:

Patient is at least 18 years of age, willing to sign and date the study PIC form and is planned to undergo at least one of the following:

1. Patient suffering from heart failure (FE<35%) undergoing de novo single or dual-chamber ICD or CRT-D system implant according to the most recent European Society of Cardiology guidelines
2. Patient suffering from heart failure (FE<35%) with a pre-existing CIED and planned to undergo ICD or CRT-D replacement or upgrading.
3. Antibiotic prophylaxis before procedure, surgical preparation with alcoholic chlorhexidine or povidone-iodine, measures to avoid pocket haematoma (avoid heparin bridging, discontinue antiplatelets if possible excluding cardioaspirin) according to current guidelines.

Exclusion Criteria:

1. Life expectancy of < 12 months or planned to undergo heart transplantation within 6 months.
2. Prior history of CIED infection, including endocarditis, in the past 12 months.
3. Clinical or laboratory sign or symptoms of active infection
4. Female patient who is pregnant, or of childbearing potential and not on a reliable form of birth control. Women of childbearing potential are required to have a negative pregnancy test within 7 days prior to device procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-06-06 (Estimated); Study Completion 2024-06-06 (Estimated)

PRIMARY OUTCOMES:
Major CIED infections occurring within Twelve months after index procedure | 12 months
  The primary study objective is to evaluate the rate of major CIED infections through 12-months post-procedure in high-risk patients.
  Major CIED infection will be defined as a device infection involving any part of the anatomy other than the incision or subcutaneous tissue, which was opened or manipulated during the CIED implantation operation, or as endocarditis defined according to the modified Duke Criteria, that resulted in CIED system removal, an invasive CIED procedure (e.g., pocket revision without removal), treatment with long-term antibiotic therapy (if the patient was not a candidate for system removal) with infection recurrence after discontinuation of antibiotic therapy, or death. CIED infections that will not meet one or more of the criteria for major infection will be classified as minor CIED infections.

SECONDARY OUTCOMES:
Adverse events after cardiac implantable electronic device implantation | 12 months
  Major mechanical complication and major and/or minor CIED infection rate throughout the duration of the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rapacciuolo, MD, PhD, Principal Investigator — Federico II, Naples
Locations (1):
- Prof Antonio Rapacciuolo,MD, PhD, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We are planning how to share IPD